CLINICAL TRIAL: NCT07400809
Title: Retrospective Cervical Cancer Oligo States (Recurrence, Metastasis) Multicentre Outcomes Study.
Acronym: Retro-COSMOS
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Dr. Supriya Sastri, Tata Memorial Hospital
Other Study IDs: TMC IEC III 900891
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chemotherapy; Treatment Compliance; Radiotherapy; Cervix Cancer; Surgery; Recurrent; Metastasis
Keywords: Recurrent and Metastatic Cervix Cancer; Oligo States
MeSH Terms: conditions — Patient Compliance; Uterine Cervical Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with oligo-recurrent and (induced) oligo-metastatic cervix cancer and treated wit: 1. Cervical cancer with (induced) oligo-metastatic and/or oligo-recurrent cervix cancer whether treated or not treated with radiation. These patients may have received previous treatment within or outside approved clinical trials/studies.
  2. Patients with poly-metastatic disease with good response to systemic chemotherapy and treated with radiation to recurrence or metastatic site.
  3. Patients treated with radical doses at the time of first diagnosis of oligo-metastasis/oligo-recurrence and present with further oligo-progression.
  4. Patients with oligo-metastasis or oligo-recurrence treated with other locally directed therapies (like surgery, ablation, etc.) are also permitted.
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable- observational study

SUMMARY:
Systemic chemotherapy with or without palliative radiation represents the current standard of care in patients with recurrent or metastatic cervix cancer. In addition, pelvic radiotherapy including brachytherapy is also recommended. There is no consensus on the treatment of metastatic site in patients with oligo-metastatic or oligo-recurrent cervix cancer. Also, it is not clear if addition of local treatment to systemic chemotherapy benefits all patients with metastatic disease or a select few with limited systemic disease burden. It's presently unclear which patients derive maximum benefit with integration of radiation at both primary and metastatic site, who develop infield recurrence if performing salvage surgery, locally directed treatments or re-irradiation in addition to systemic chemotherapy improves overall outcomes. The heterogeneity in clinical practice provides an important opportunity to develop a framework for data collection and future studies within such subgroup of patients. In this retrospective study, we aim to determine overall survival, Infield progression free survival, overall progression free survival, dose response relationship of nodal and visceral progressions, and within setting of re-irradiation (infield progressions), severe adverse events and toxicity, risk groups identification, a nomogram which correlates risk groups with expected outcomes, and framework for tissue collection for translational research Investigators will record the parameters in a predesigned proforma without including personal identifiers.

DETAILED DESCRIPTION:
This is a multicentric, retrospective registry designed to evaluate clinical outcomes in patients with (induced) oligo-metastatic and oligo-recurrent cervical cancer. These patients will be identified using an adapted ESTRO-ASTRO consensus definition. The study aims to investigate the role of radiation therapy-whether high-dose, stereotactic ablative, or re-irradiation-in combination with or without systemic chemotherapy, immunotherapy, or targeted agents, in improving survival outcomes and minimizing treatment-related toxicity. Despite systemic chemotherapy being the current standard for metastatic cervical cancer, the survival benefits remain modest. Emerging evidence, including findings from the SABR-COMET trial and institutional experiences, suggests that selected patients with limited metastatic burden may derive survival benefit from integration of local therapies. However, for cervical cancer specifically, there is limited consensus on the optimal use of radiation in the oligometastatic or oligorecurrent setting.

This registry seeks to capture real-world data from EMBRACE-participating centers to explore treatment patterns, dose-response relationships, and toxicity profiles. The primary objective is to determine overall survival, with secondary endpoints including in-field and overall progression-free survival, treatment-related toxicity, and development of prognostic risk groups. The registry will also support development of a nomogram and a framework for future translational research, including tissue collection. Data will be collected through a centralized, secure electronic data capture system (Castor EDC) hosted at Erasmus University Medical Center. Each participating site will enter anonymized patient data into standardized case report forms derived from patient records. Built-in data validation rules and consistency checks will be used to ensure data quality, with each center responsible for accuracy and source verification. A central data dictionary standardizes variable definitions and coding. The data will be managed under established standard operating procedures covering data collection, quality control, and analysis. Statistical analysis will include descriptive summaries, Kaplan-Meier survival curves, Cox regression modeling, and dose-response assessments. Approximately 350-400 patients treated between 2007 and 2021 are expected to be included. The registry does not involve direct patient contact and poses minimal risk, with all ethical approvals and data protection safeguards in place, including local IRB clearance and waiver of consent where applicable. This registry aims to inform future clinical trials and guidelines for personalized treatment in oligo-metastatic and oligo-recurrent cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical cancer with (induced) oligo-metastatic and/or oligo-recurrent cervix cancer whether treated or not treated with radiation. These patients may have received previous treatment within or outside approved clinical trials/studies.
2. Patients with poly-metastatic disease with good response to systemic chemotherapy and treated with radiation to recurrence or metastatic site.
3. Patients treated with radical doses at the time of first diagnosis of oligo-metastasis/oligo-recurrence and present with further oligo-progression.
4. Patients with oligo-metastasis or oligo-recurrence treated with other locally directed therapies (like surgery, ablation, etc.) are also permitted.

Exclusion Criteria:

1. Gynaecological cancer other than cervical cancer.
2. Persistent Poly-metastatic disease post systemic treatment
3. Receiving investigational new drugs at the time of relapse as part of other ongoing trials.
4. No clinical follow up after treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We aim to include all patients with (induced) oligo metastatic and oligo recurrent setting irrespective whether radiation was used or not with an aim to have different cohorts of patients based on interventions used. This will allow to better understand outcomes and radiation dose response if any. Also this provides an opportunity to better understand impact of radiation potentially through a matched pair analysis in future.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2027-06-14 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 4 years
  To determine the overall survival (OS) of patients diagnosed with oligo-recurrent and (induced) oligo-metastatic cervical cancer treated with radiation or other local therapies, with or without systemic chemotherapy. Overall survival is defined as the time from registration to death from any cause or the last follow-up.

SECONDARY OUTCOMES:
Infield Progression-Free Survival (PFS) | 4 years
  Time from registration to progression of disease within the treated radiation or local therapy field, death from any cause, or last follow-up.
Overall Progression-Free Survival (PFS) | 4 years
  Time from registration to any disease progression (local, regional, or distant), death from any cause, or last follow-up.
Dose-Response Relationship of Nodal and Visceral Progressions | 4 years
  Evaluation of the relationship between radiation dose delivered and subsequent progression in nodal and visceral sites, with outcomes measured as time from registration to progression at these specific sites, death from any cause, or last follow-up.
Dose-Response Relationship in Re-irradiation Settings | 4 years
  Assessment of the correlation between radiation dose and infield progression in patients undergoing re-irradiation, measuring time to progression, death, or last follow-up.
Severe Adverse Events and Toxicity | 4 years
  Evaluation and documentation of grade ≥3 treatment-related adverse events and toxicities occurring during or after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Supriya Chopra, MD, Principal Investigator — ACTREC, Tata Memorial Centre, Navi Mumbai India
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided